CLINICAL TRIAL: NCT03983317
Title: Pilot Evaluation of the Empower Neuromodulation System in Alcohol Use Disorder (AUD) Patients
Brief Title: Pilot Evaluation of the Empower Neuromodulation System in AUD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRD-12-1176-01; R43AA027188-01 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: All participants will have a one-week control period with no treatment followed by two weeks of twice daily Empower treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Baseline (No Intervention): For the first week of the study, participants will not administer treatment with the Empower device. Participants will complete surveys to establish baseline values for each participant.
- Active treatment (Experimental): Participants will self-administer treatment with the Empower device two times daily for two weeks. Participants will complete surveys over the two-week period to evaluate the effects of the Empower treatment.
  Interventions: Device: Empower Neuromodulation System

INTERVENTIONS:
Device: Empower Neuromodulation System — Transcutaneous electrical nerve stimulation
  Arms: Active treatment

SUMMARY:
This study evaluates the effects of peripheral nerve stimulation on alcohol craving and consumption in participants with alcohol use disorder (AUD). This is a pilot investigation in which all participants will receive the active treatment.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a major public health concern, affecting over 16 million Americans. Peripheral nerve stimulation via acupuncture has been shown to directly decrease alcohol craving and self-administration. TheraNova has developed the Empower Neuromodulation System, a non-invasive, portable transcutaneous electrical nerve stimulation (TENS) device intended to stimulate peripheral nerves for the treatment of AUD. In this study, we will conduct a cross-over, home-use study in participants with AUD. Participants will have a one-week control period with no treatment followed by two weeks of twice daily treatment with the Empower device. We will evaluate endpoints for safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 21 year of age at Visit 1
* Has a current diagnosis of alcohol use disorder per DSM-5 by clinician assessment
* Endorses Criterion 4 in DSM-5
* Has a desire to maintain abstinence or, if not abstinent, a desire to reduce or quit alcohol use
* Has a breath alcohol concentration of 0.00% at enrollment
* Is able to provide informed consent
* Is able to understand spoken and written English
* Is capable and willing to follow all study-related procedures

Exclusion Criteria:

* Has been diagnosed with unstable psychosis, epilepsy, peripheral neuropathy, or nerve damage
* Requires acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD)
* Has implanted electrical and/or neurostimulator device (e.g. pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
* Has an electrically conductive metal object (e.g. jewelry) that cannot be removed from the palm and will directly contact the gel electrodes of the Empower Neuromodulation System
* Will not, for the duration of the participation in the study, have a living situation that provides regular access to an electrical outlet.
* Is pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Has used an investigational drug/device therapy within the past 4 weeks
* Is deemed unsuitable for enrollment in the study by the PI

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jaasma, Study Director — Theranova, L.L.C.
Locations (1):
- NCIRE, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the Baseline Phase first, so participants who did not complete the Baseline Phase did not start the Treatment Phase.
Groups:
- Active Treatment: For the first week of the study, participants did not administer treatment with the Empower device. In this one-week Baseline Phase, participants only completed surveys to establish baseline values. In the final two weeks of the study, participants self-administered treatment with the Empower device two times daily. Participants completed surveys over the two-week period to evaluate the effects of the Empower treatment.
  Empower Neuromodulation System: Transcutaneous electrical nerve stimulation
Period: Overall Study
Arm/Group | Active Treatment
Started | 25
Completed | 20
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 58 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 11
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Alcoholic Drinks Consumed Per Day
Description: Change in the self-reported average daily consumption over the final week (Week 2) of the treatment phase compared to the week of the pre-treatment baseline phase.
Time Frame: Baseline week and Week 2 of the treatment phase
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: Change in alcoholic drinks per day
Arm/Group | Active Treatment
Number analyzed (Participants) | 20
Change in alcoholic drinks per day | -1.1 (1.7)
Statistical Analysis 1: Comparison: Active Treatment; Test type: Other — We tested if the average drinks consumed was statistically different in Week 2 of the Treatment Phase vs. the Baseline Phase. This was evaluated via a paired t-test; p = 0.026, t-test, 2 sided; Paired t-test

2. Primary Outcome: Number of Participants With Adverse Events
Description: Safety assessment via device-related adverse events
Time Frame: Through study completion, an average of 3 weeks
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Decrease in Mean Alcohol Craving Intensity
Description: Change in self-reported average alcohol craving intensity via 100-mm visual-analog scale (VAS). The VAS has a minimum score of 0 (no craving) and a maximum score of 100 (severe craving). We compared the average daily craving intensity over the final week (Week 2) of the treatment phase compared to the week of the pre-treatment baseline phase.
Time Frame: Baseline week and Week 2 of the treatment phase
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: Change in units on 100-mm VAS scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 20
Change in units on 100-mm VAS scale | -13 (17)
Statistical Analysis 1: Comparison: Active Treatment; Test type: Other — We tested if the average craving intensity was statistically different in Week 2 of the Treatment Phase vs. the Baseline Phase. This was evaluated via a paired t-test; p = 0.001, t-test, 2 sided; Paired t-test

4. Secondary Outcome: Usability
Description: System Usability Scale (SUS) survey to evaluate usability. The SUS is a 10-item self-report survey (each question is answered on a 5-point Likert scale) which measures usability. An SUS score of 68 is considered average, whereas SUS=80 is the 90th percentile score ("excellent").
Time Frame: Study completion, at approximately 3 weeks
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: Score on the SUS survey scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 20
Score on the SUS survey scale | 76 (15)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Active Treatment (AEs Occurred During the Two-week Treatment Phase): For the first week of the study, participants did not administer treatment with the Empower device. In this one-week Baseline Phase, participants only completed surveys to establish baseline values. In the final two weeks of the study, participants self-administered treatment with the Empower device two times daily. Participants completed surveys over the two-week period to evaluate the effects of the Empower treatment.
  Empower Neuromodulation System: Transcutaneous electrical nerve stimulation
Arm/Group | Active Treatment (AEs Occurred During the Two-week Treatment Phase)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (AEs Occurred During the Two-week Treatment Phase) (N=25)
Deep vein thrombosis (Vascular disorders) | 1 (1) — Determined to not be device-related
Head injury (General disorders) | 1 (1) — Slip/fall with head injury. Determined to not be device-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03983317/Prot_SAP_000.pdf